CLINICAL TRIAL: NCT04629690
Title: The Impact of Frailty Screening of Older Adults With muLtidisciplinary Assessment of Those At Risk During Emergency Hospital Attendance on the Quality, Safety and Cost-effectiveness of Care (SOLAR): a Randomised Controlled Trial
Brief Title: SOLAR- Frailty Screening and Multidisciplinary Assessment of Older Adults in the Emergency Department
Acronym: SOLAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Collaborators: University Hospital of Limerick (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOLAR
Record Dates: First submitted 2020-11-02; First posted 2020-11-16 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Frailty
Keywords: Comprehensive Geriatric Assessment; Emergency Department; Older Adults; Frailty
MeSH Terms: conditions — Frailty; Emergencies | interventions — Geriatric Assessment

STUDY DESIGN:
Intervention Model Description: Randomised control trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be unaware if the participant was in control or intervention arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): The control group will obtain usual medical care in the Emergency Department and Acute Medical Assessment Unit
- SOLAR arm (Experimental): The SOLAR arm will obtain a comprehensive geriatric assessment which will be provided by a geriatric doctor, physiotherapist, occupational therapist, social worker, pharmacist and specialist nurse.
  Interventions: Other: SOLAR

INTERVENTIONS:
Other: SOLAR — The participants will obtain a multidisciplinary assessment regarding their medical conditions, medication review, cognitive assessment, functional assessment, gait and balance assessment by senior clinicians and a management plan will be implemented.
  Other Names: Comprehensive Geriatric Assessment
  Arms: SOLAR arm

SUMMARY:
SOLAR is a randomised control trial exploring the role of Comprehensive Geriatric Assessment (CGA) in older adults who screen positive for frailty based on the Identification of Seniors at Risk (ISAR) tool the the Emergency Department and Acute Medical Assessment Unit of a University Teaching Hospital.

DETAILED DESCRIPTION:
All patients who are over seventy-five will be screened for frailty using the widely used ISAR tool. Those with a score of 2 or above in the ISAR will be randomised. The treatment arm will undergo geriatric medicine team-directed CGA from admission to Emergency Department (ED) or Acute Medical Assessment Unit (AMAU) whereby the non-treatment arm will undergo usual patient care. A dedicated multidisciplinary team of a geriatric medicine trainee, physiotherapist, occupational therapist and medical social worker will carry out the assessment, as well as interventions that arise from that assessment. Primary outcomes will be time from triage to decision to admit or discharge. Secondary Outcomes will be subsequent Emergency Department reattendance, rehospitalisation, functional decline and mortality at 30 days and 180 days. This will be recorded by telephone consultation and electronic records.

ELIGIBILITY:
Inclusion Criteria:

* Older adults aged 75 years or over
* Medically stable as deemed by the treating physician
* A score of 2 or above on the ISAR
* Present with a medical complaint

Exclusion Criteria:

* Those under the age of 75 years
* A score of less than 2 on the ISAR
* Acute myocardial infarction, stroke or non-medical problems e.g. surgical or psychiatric issues
* Patients who are medically unstable
* If neither the patient nor carer can communicate in English sufficiently to complete consent or baseline assessment
* Confirmed or highly suspicious of symptoms for COVID 19.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 229 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Patient Experience Times (PET) | Exact time of admission or discharge from ED will be collected at 30 days from index visit
  PET time recorded as time of arrival at the ED to discharge or admission
Time to admission or discharge and if for admission, time that the bed is booked to go to medical wards. | Exact time of admission or discharge from ED will be collected at 30 days from index visit
  This is the time that the patient is either discharged or identified for admission and bed booked to go to the medical wards

SECONDARY OUTCOMES:
Rate of ED Representation | 30 days and 6 months
  A record of the patient coming back to the ED within 30 days and/or 6 months
Mortality | 30 days and 6 months
  A record of the patient having died within 30 days or 6 months
Rate of Hospital Readmission | 30 days and 6 months
  A record of the patient requiring admission to the hospital within 30 days or 6 months
Functional Decline | 30 days and 6 months
  As determined by the Barthel Index. Barthel Index is a score from 0-20. A score of 0 is completely dependent, 20 is fully independent.
Patient Satisfaction- | 30 days
  As determined by the Patient Satisfaction Survey III Short Form (PSQ18). This is scored from 18 to 90. 18 being the worst score and 90 being the best score.
Patient Quality of Life | 30 days
  As determined by the Euro Quality of Life (Qol) EQ5D. Scored from 0 to 100. 0 is worst imaginable health state with 100 being the best imaginable health state
Number of visits to family doctor, therapists or public health nurse | 30 days and 6 months
  Determined by self reported visits to family doctor, allied health services or Public Health Nurse. There will be a telephone consultation at 30 days and 6 months where patients will be asked if they have visited a family doctor, therapist or public health nurse in the previous 30 days at the 30 day telephone call, or 6 months at the 6 month phone call.

CONTACTS AND LOCATIONS:
Overall Officials: Rose Galvin, phD, Principal Investigator — University of Limerick
Locations (1):
- University Hospital Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Individual data will be stored on a data repository after the study analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The study protocol will be prepared for publication in an open access journal. the study protocol will include the Statistical Analysis Plan and Informed Consent Form. It is likely to be published in Quarter 2 of 2021.
  The Clinical Study Report will be made publicly available in the form of a peer reviewed publication in late 2021.
Access Criteria: Supporting information will be available on peer reviewed publications.

REFERENCES:
- [Background] McCusker J, Bellavance F, Cardin S, Trepanier S, Verdon J, Ardman O. Detection of older people at increased risk of adverse health outcomes after an emergency visit: the ISAR screening tool. J Am Geriatr Soc. 1999 Oct;47(10):1229-37. doi: 10.1111/j.1532-5415.1999.tb05204.x. PMID 10522957
- [Derived] Leahy A, Barry L, Corey G, Whiston A, Purtill H; SOLAR team; Shanahan E, Shchetkovsky D, Ryan D, O'Loughlin M, O'Connor M, Galvin R. Frailty screening with comprehensive geriatrician-led multidisciplinary assessment for older adults during emergency hospital attendance in Ireland (SOLAR): a randomised controlled trial. Lancet Healthy Longev. 2024 Nov;5(11):100642. doi: 10.1016/j.lanhl.2024.100642. Epub 2024 Nov 11. PMID 39541993
- [Derived] Leahy A, McNamara R, Reddin C, Corey G, Carroll I; SOLAR team; O'Neill A, Flannery D, Devlin C, Barry L, MacCarthy B, Cummins N, Shanahan E, Shchetkovsky D, Ryan D, O'Connor M, Galvin R. The impact of frailty Screening of Older adults with muLtidisciplinary assessment of those At Risk during emergency hospital attendance on the quality, safety and cost-effectiveness of care (SOLAR): a randomised controlled trial. Trials. 2021 Aug 31;22(1):581. doi: 10.1186/s13063-021-05525-w. PMID 34465368